CLINICAL TRIAL: NCT03740269
Title: Oral Health Educational Program for Knowledge, Attitude and Practice (KAP) of Oral Health Among a Group of Egyptian School Girls in Ras Sedr - South Sinai
Brief Title: Oral Health Educational Program for Knowledge,Attitude,Practice of Oral Health Among Agroup of Egyptian School Girls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rana Abd El-Sattar Omar Ramadan (Other)
Responsible Party: Sponsor-Investigator, Rana Abd El-Sattar Omar Ramadan, postgraduate student in Faculty of Dentistry Cairo university, Cairo University
Organization: Cairo University (Other)
Other Study IDs: CEBD-CU-2018-07-04
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: oral health education; oral health promotion; oral health education program; oral hygiene status; knowledge,attitude,practice; oral health knowledge,attitude,practice; oral hygiene knowledge,attitude,practice; knowledge,attitude,practice oral health; knowledge,attitude,practice oral hygiene; KAP
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oral health educational program: poster for oral health education program for a group of egyptian school girls
  Interventions: Other: oral health educational program

INTERVENTIONS:
Other: oral health educational program — poster education about the important of oral health status, different brushing technique, different tooth paste, the balanced diet, changes occur to their mouth during the puberty period

SUMMARY:
This study will demonstrate oral health educational program to egyptian school girls age from 12-14 years old to evaluate the change in the knowledge, attitude and practice of oral health

DETAILED DESCRIPTION:
According to World Dental Federation 2017 oral health is defined as multi-faceted and include the ability to speak, smile, smell, taste, chew, swallow, and convey a range of emotions through facial expressions with confidence and without pain, discomfort, and disease of the craniofacial complex .Oral disease constitute a significant public health problem in developing countries due to their high prevalence, economic consequence and negative impact on the quality of the life of affected individual.

Estrogen cause change in the blood vessels and progesterone stimulate the production of inflammatory mediators which lead to increase of gingival inflammation appear as gingival enlargement, increase in gingival bleeding and crevicular fluid flow and microbial changes.

The oral health education is important tool to make the primary level of prevention. So the benefits from health education is to improve knowledge and awareness of children which results on developing favorable oral behavior and so favorable oral health status.

.As the school is consider a place for gathering large number of children so it is ideal place for conducing successful health education.

this study will Identify baseline oral hygiene knowledge, attitude and practice among 12-14 years old school children. then Record oral hygiene status by oral hygiene index simplified after that assess the effectiveness of oral health education in modifying oral health knowledge, attitude and practice

ELIGIBILITY:
Inclusion Criteria:

* girls age 12 - 14 years old

Exclusion Criteria:

* refusal to participate in the research

Ages: 12 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: consecutive convenient sampling recruiting all girls attending the school in that day
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
knowledge, attitude and practice of oral health | 3 months
  self reported questionnaire for knowledge, attitude and practice before and after oral health educational program
oral hygiene index simplified | 3 months
  record amount of plaque and calculus accumulation before and after oral health educational program

CONTACTS AND LOCATIONS:
Overall Officials: hassan ahmed, Principal Investigator — center of evidence based dentistry

IPD SHARING:
Plan to Share IPD: Undecided
due to financial issue